CLINICAL TRIAL: NCT03531671
Title: The Future of Cataract Assessment: Investigation of the Utility of a Novel Binocular OCT System for Clinical Application
Brief Title: Assessing the Optics of the Eye Pre- and Post-operatively in Cataract
Acronym: CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: KEAP1003
Record Dates: First submitted 2018-03-13; First posted 2018-05-22 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Assessing age related cataract, all 200 subjects will have whole eye OCT scan performed during their pre-operative cataract assessment and 50 subjects (all subjects requested to participate until 50 subject criteria met) will have these assessments reassessed during their post-operative assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Presence of age related cataract (Experimental): Binocular-OCT used to assess the eye pre and post-operatively.
  Interventions: Device: Binocular-OCT

INTERVENTIONS:
Device: Binocular-OCT — Binocular Optical Coherence Tomographer used to assess both eyes in the same session without the need for a trained assistant.

SUMMARY:
The purpose of the study is to investigate if a novel instrument called a Binocular Optical Coherence Tomographer (OCT) may resolve many of the issues with the assessment of patients with cataract.

DETAILED DESCRIPTION:
Cataract is the second leading cause of blindness in western Europe but the leading cause of blindness in the developing world and both central and eastern Europe. The most common cause of cataract is age. A number of clinical assessments are required to assess the status and suitability of each patient for cataract surgery. Currently, these procedures are performed in an inefficient manner with the patient having to move to different clinical areas to access often large instruments that are costly to both purchase and maintain. Such an inefficient patient pathway has been identified as a factor that can markedly increase the cost of outpatient appointments, extend waiting times, and crucially lead to a reduction in patient satisfaction. A novel instrument that offers a solution to such problems is the recently developed Binocular Optical Coherence Tomographer. Binocular-OCT is capable of non-invasively imaging the whole-eye in a potentially small, inexpensive and portable device and is also capable of capturing images from both eyes in the same session without the need for assistance from a trained technician. The Binocular-OCT has the capability to perform the functions of many clinical tools in a single instrument. Of particular relevance to the assessment of the patient with cataract is the ability to capture high resolution images of the anterior eye and crystalline lens with swept-source OCT technology. In this study, the proposed advantages of binocular OCT system will be assessed for the management of cataract.

This research is important, to not only improve cataract assessment and optomise surgical outcomes, but it is also vital to establish sensitive measures of lens quality to determine tools to aid trails attempting to retard the progression of cataract.

ELIGIBILITY:
Inclusion Criteria:

* - Presence of cataract
* Male or female, aged 18 years or older
* Ability to understand nature/purpose of the study and to provide informed consent
* Ability to undergo binocular OCT imaging
* Ability to follow instructions and complete the study
* Ability to speak English

Exclusion Criteria:

* - Hearing impairment sufficient to interfere with hearing instructions
* Any condition which, in the investigator's opinion, would conflict or otherwise prevent the subject from complying with the required procedures, schedule, or other study conduct.
* Any cases where the globe has been affected by trauma, etc.
* Traumatic aetiologies of cataract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Feasibility | 18 Months
  Investigate the feasibility of the Binocular-OCT to produce accurate biometric measurements of the eye, via calculation of quantitative cataract density and localisation index from the binocular-OCT image of the lens.

SECONDARY OUTCOMES:
Post-Operative Measurements | 18 Months
  Examining the ability of the Binocular-OCT to perform post-operative assessments of the lens position.
Post-Operative Measurements | 18 Months
  Examining the ability of the Binocular-OCT to perform post-operative assessments of the ocular clarity.
Post-Operative Measurements | 18 Months
  Examining the ability of the Binocular-OCT to perform post-operative assessments of the retinal thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Pearse Keane, Study Director — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data retained within the central research team.